CLINICAL TRIAL: NCT03174340
Title: Evaluation of Exercise, in Addition to Diet, in Women With Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Michel Boulvain, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-080 MATPED 07-021
Record Dates: First submitted 2017-01-24; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + diet (Experimental): Exercise intervention:
  During the first session a standardized exercise prescription will be discussed with the participant. The exercise program will be of a moderate intensity, at less than 140 heart beats/min (which corresponds to 60% of the calculated maximum heart rate (HRmax) or 50% maximum oxygen volume (VO2max) ). A session of 30 to 60 minutes/week will be organised.
  * Participants will be instructed to conduct a nonsedentary lifestyle. They will be encouraged to increase their number of steps on a daily basis and perform not more that 45 minutes of continuous exercise per day. Pedometers will be used to measure the compliance and as a positive feedback for motivation.
  * The participants will return to the exercise laboratory once per week for Actiheart data downloading, number of steps recording, exercise support and counselling, and to perform the supervised group exercise intervention.
  This is in addition to the diet (see below, control group)
  Interventions: Behavioral: Exercise
- Diet only (No Intervention): Participants will receive diet counselling according to their characteristics. The usual recommendation is to have a fractioned normocaloric diet (unless the dietician identify a grossly hypercaloric diet), with low fat and increase in fibers content.

INTERVENTIONS:
Behavioral: Exercise — Once per week, participants will be enrolled in supervised group exercise intervention. They will be encouraged in walking 45 minutes per day
  Arms: Exercise + diet

SUMMARY:
The main objective is to evaluate the effect of therapeutic exercise program on blood glucose regulation in women with gestational diabetes mellitus (GDM) who are assigned to diet-and-exercise, compared to diet only (usual treatment). The primary outcome is the need for insulin treatment in the two groups.

DETAILED DESCRIPTION:
In women with gestational diabetes, light to moderate daily physical activity may a useful therapeutic approach to improve the control of glycaemia and decrease the need for prescription of insulin. Increased physical activity in pregnant women with gestational diabetes is expected to decrease the mother and child morbidity associated with gestational diabetes, but also to improve the general health status of the mother and the child.

The objectives of this randomized trial are:

* To evaluate the effect of therapeutic exercise program on blood glucose regulation in women with GDM who are assigned to diet-and-exercise protocol.
* To demonstrate the feasibility of the therapeutic exercise treatment and the possibility of using the exercise program as an optional therapeutic approach for women with GDM.

ELIGIBILITY:
Inclusion Criteria:

* gestational diabetes, based on the criteria of Coustan-Carpenter, then on the International Association Diabetes Pregnancy Study Groups (IADPSG )

Exclusion Criteria:

* pre-existing diabetes
* twins

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2008-02-21 (Actual); Primary Completion 2013-04-25 (Actual); Study Completion 2013-06-19 (Actual)

PRIMARY OUTCOMES:
Prescription of insulin during the follow-up | From inclusion in the study (randomization usually between 24 and 30 weeks of gestation) until the end of pregnancy (delivery, usually 38 to 41 weeks of gestation). It is impossible in our context to give a specific time point.
  The primary outcome will include any amount (dosage) of insulin and any frequency of injection. Prescription of insulin is considered when glycaemia is above 5.3 mmol/L fasting and/or above 8.0 at 1 hour after the meal.

SECONDARY OUTCOMES:
Control of glycemia | From inclusion in the study (randomization usually between 24 and 30 weeks of gestation) until the end of pregnancy (delivery).
  4 times per day, participants will check their blood sugar level. The investigators will record these blood sugar levels and consider as normal if below 5.3 mmol/L fasting and below 8.0 at 1 hour after the meal. Suboptimal glycemic control will be defined as 2 or more glycemia above these target values; good control will be defined as less than 2 values above the thresholds. The variable "good glycemic control" will be coded "yes" if the above criteria (<2 abnormal values) are met, and "no" otherwise (>=2 abnormal values)
Compliance with the exercise (in the exercise group only) | From inclusion in the study (randomization usually between 24 and 30 weeks of gestation) until the end of pregnancy (delivery).
  Satisfactory compliance will be defined as walking at least 5000 steps/day 5 days a week and attending at 50% or more of the weekly supervised exercise program. The variable "compliance" will be coded "yes" if both the above criteria are met, and "no" otherwise

OTHER OUTCOMES:
Timing of insulin treatment | From inclusion in the study (randomization usually between 24 and 30 weeks of gestation) until the end of pregnancy (delivery).
  To better understand the effect of the intervention on the primary outcome, prescription of insulin), the investigators will compare between groups:
  Time between randomization and insulin prescription (days)
Gestational age at start of insulin treatment | From inclusion in the study (randomization usually between 24 and 30 weeks of gestation) until the end of pregnancy (delivery).
  the investigators will compare between groups: Gestational age at start of insulin treatment (weeks) (mean ± SD)
Dosage of long-acting insulin | From inclusion in the study (randomization usually between 24 and 30 weeks of gestation) until the end of pregnancy (delivery).
  Maximal dose of long-acting insulin per day (mean ± SD)
Dosage of short-acting insulin | usually between 24 and 30 weeks of gestation) until the end of pregnancy (delivery).
  Maximal dose of short-acting insulin per day (mean ± SD)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Boulvain, Principal Investigator — University Hospital, Geneva

IPD SHARING:
Plan to Share IPD: Yes
Meta-analysis with the Cochrane Collaboration, if individual patient data are needed

REFERENCES:
- [Derived] Boulvain M, Othenin-Girard V, Jornayvaz FR, Kayser B. Impact of an exercise program combined with dietary advice on avoiding insulin prescription in women with gestational diabetes: a randomized controlled trial. Diabetol Metab Syndr. 2024 Sep 30;16(1):238. doi: 10.1186/s13098-024-01470-1. PMID 39343942